CLINICAL TRIAL: NCT00086619
Title: Evaluation of Factors That Affect Skeletal Responses to PTH
Brief Title: Parathyroid Hormone (PTH) for Osteoporosis in Postmenopausal Women
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: National Institute of Arthritis and Musculoskeletal and Skin Diseases (NIAMS) (NIH)
Responsible Party: Principal Investigator, Robert M. Neer, MD, Associate Professor of Medicine, Massachusetts General Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NIAMS-123; 1P50AR044855 (NIH)
Record Dates: First submitted 2004-07-07; First posted 2004-07-08 (Estimated); Results first posted 2013-09-26 (Estimated); Last update posted 2013-10-30 (Estimated); Status verified 2013-09

CONDITIONS: Postmenopausal Osteoporosis; Osteoporosis
Keywords: Osteoporosis; Parathyroid hormone; Teriparatide; Bone formation; Bone resorption
MeSH Terms: conditions — Osteoporosis, Postmenopausal; Osteoporosis; Bone Resorption

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- constant dose (Experimental): Participants will receive synthetic human parathyroid hormone fragment 1-34 (hPTH 1-34) once-daily in a constant dose of 30 mcg/day.
  Interventions: Drug: synthetic hPTH 1-34
- ascending dose (Experimental): Participants will receive synthetic human parathyroid hormone fragment 1-34 (hPTH 1-34) once-daily in a dose that ascends at 6 month intervals (20-30-40 mcg/day).
  Interventions: Drug: synthetic hPTH 1-34

INTERVENTIONS:
Drug: synthetic hPTH 1-34 — Either daily treatment with self-injected hPTH 1-34 or ascending dose treatment at 6-month intervals of hPTH 1-34
  Other Names: synthetic human parathyroid hormone 1-34

SUMMARY:
Parathyroid hormone (PTH) increases bone formation and thereby improves bone density and bone strength in postmenopausal women with osteoporosis. However, prolonged PTH treatment increases bone formation less and less over time. This study will test whether increasing the daily dose of PTH sustains its ability to improve bone formation, and optional sub-studies will test several potential reasons why PTH's effects on bone formation decline over time.

DETAILED DESCRIPTION:
In women with postmenopausal osteoporosis, PTH increases bone mineral density more than anti-resorptive agents, and its use markedly reduces the incidence of new spine and non-spine fractures. Still, PTH is not a cure for osteoporosis in many patients because PTH-stimulated bone formation declines as PTH therapy continues. Biochemical analyses suggest that bone formation and resorption peak after 6 to 9 months of daily PTH therapy and then decline progressively.

The study will last 18 months. Blood, urine, and bone density tests will occur at screening. At the start of the study, participants will be randomly assigned to one of two PTH dose regimens. Patients will go to Massachusetts General Hospital at Months 0, 3, 6, 9, 12, 15, and 18 for blood and urine collection. In addition, bone density tests by DXA will be performed at Months 0, 6, 12, and 18, and by quantitative CT scans at Months 0 and 18. Approximately 6 weeks after any change in PTH dose, each participant's blood calcium will be checked 4 to 6 hours after that day's PTH injection, and her 24-hour urine calcium excretion will also be checked.

Participants may enroll in optional substudies that will test whether reduced skeletal responses to long-term treatment with PTH are accompanied by changes in its absorption and/or destruction and whether reduced skeletal responses to long-term treatment with PTH are accompanied by parallel reductions in kidney responses to PTH.

ELIGIBILITY:
Inclusion Criteria:

* Three or more years after menopause
* Bone mineral density T-score < or = -2.0 by dual-energy x-ray absorptiometry (DXA) of vertebrae or femoral neck, or by quantitative computerized tomography (QCT) of vertebral body trabeculae

Exclusion Criteria:

* Cannot walk without assistance
* Significant heart, kidney, liver, or malignant disease
* Current alcohol abuse
* Major psychiatric disorders
* Other current or past disorders known to affect bone
* Use of medications known to affect bone for > 7 days in the past 12 months
* Use of bisphosphonates or fluoride
* Abnormal blood calcium, PTH, 25-hydroxy vitamin D, creatinine, liver function tests, or complete blood count
* Elevated calcium levels in 24-hour urine collection

Ages: 46 Years to 85 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2004-05; Primary Completion 2009-12 (Actual); Study Completion 2009-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robert M. Neer, MD, Principal Investigator — Massachusetts General Hospital; Joel S. Finkelstein, MD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

REFERENCES:
- [Result] Yu EW, Neer RM, Lee H, Wyland JJ, de la Paz AV, Davis MC, Okazaki M, Finkelstein JS. Time-dependent changes in skeletal response to teriparatide: escalating vs. constant dose teriparatide (PTH 1-34) in osteoporotic women. Bone. 2011 Apr 1;48(4):713-9. doi: 10.1016/j.bone.2010.11.012. Epub 2010 Nov 24. PMID 21111078

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Postmenopausal women with low bone density were recruited from 2004-2007 to participate in this study at a single academic medical center. Recruitment letters were sent to women in the Greater Boston area and the trial was also posted on clinicaltrials.gov.
Pre-assignment Details: Must satisfy inclusion and exclusion criteria.
Groups:
- Constant Dose PTH: Participants received constant dose synthetic hPTH 1-34 (30 mcg/day).
- Ascending Dose PTH: Participants received ascending dose synthetic hPTH 1-34 (20-30-40 mcg/day).
Period: Overall Study
Arm/Group | Constant Dose PTH | Ascending Dose PTH
Started | 40 | 40
Completed Baseline Visit | 34 | 36
Completed 12 Month Visit | 26 | 26
Completed | 25 | 23
Not Completed | 15 | 17
Not completed — Withdrawal by Subject | 6 | 6
Not completed — Adverse Event | 8 | 10
Not completed — Protocol Violation | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Constant Dose PTH | Ascending Dose PTH | Total
Number analyzed (Participants) | 40 | 40 | 80
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 26 | 27 | 53
  >=65 years | 14 | 13 | 27
Age Continuous [Mean (Standard Deviation); unit: years] | 63.3 (7.6) | 62.1 (8.9) | 62.7 (8.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 40 | 40 | 80
  Male | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 40 | 40 | 80

OUTCOME MEASURES:

1. Primary Outcome: Changes in Indices of Bone Turnover
Description: Change from month 0 (pre-treatment) baseline serum aminoterminal propeptide of type I collagen (PINP), osteocalcin (OC), and C-terminal telopeptide (CTX), expressed as an area under the curve (AUC). Each marker measurement result was multiplied by the corresponding subject-specific elapsed study time interval using the trapezoidal rule, and these products were summed to generate a subject-specific AUC (months*ng/ml) for the marker.
Time Frame: Each index of bone turnover was measured at study month 0, 1.5, 3, 6, 7.5, 9, 12, 13.5, 15, and 18.
Population: Because this was a physiologic study evaluating the impact of stepwise increases in teriparatide, per protocol analysis was performed as was pre-specified in our analysis plan. Outcomes data were analyzed in women who remained on teriparatide throughout the first stepwise increase (i.e. until month 12 or later).
Measure: Mean (Standard Deviation); unit: months*(ng/ml - baseline ng/ml)
Arm/Group | Constant Dose PTH | Ascending Dose PTH
Number analyzed (Participants) | 26 | 26
months*(ng/ml - baseline ng/ml)
  PINP | 4418 (2732) | 3696 (1735)
  OC | 956 (416) | 822 (312)
  CTX | 22 (11) | 19 (9)

2. Secondary Outcome: Change in Bone Mineral Density (BMD)
Description: Percent change in BMD of the spine, femur, radius, and ulna, and subtotal body, calculated as 100*[(final - month 0)/month 0] in subjects who took study therapy for at least 12 months.
Time Frame: baseline and 18 months (12 months in 4 subjects)
Population: Final BMD was measured after 18 months of study therapy in 48 subjects and measured after 12 months of study therapy in 4 others who thereafter dropped out prematurely. Of the latter 4, 3 were in the ascending dose arm and 1 was in the constant dose arm.
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Constant Dose PTH | Ascending Dose PTH
Number analyzed (Participants) | 26 | 26
percent change
  1/3 Radius BMD | -4.6 (2.8) | -3.1 (3.3)
  Femoral neck BMD | 1.7 (3.0) | 3.5 (2.7)
  Spine BMD | 5.9 (4.6) | 7.4 (3.8)
  Subtotal BMD | -1.6 (0.8) | -0.9 (0.5)
  Total hip BMD | 1.4 (3.1) | 1.3 (2.5)

ADVERSE EVENTS:
Arm/Group | Constant Dose PTH | Ascending Dose PTH
Serious Adverse Events (participants affected / at risk) | 0/40 | 2/40
Other Adverse Events (participants affected / at risk) | 5/40 | 8/40
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Constant Dose PTH (N=40) | Ascending Dose PTH (N=40)
Hypercalcemia requiring emergency room visit (Endocrine disorders) | 0 (0) | 1 (1) — Patient had symptoms of weakness/nausea and was found to have hypercalcemia (calcium 14.1 mg/dL). Her PTH therapy was discontinued and she was treated with IV fluids and calcitonin, resulting in normalization of calcium to 8.5 mg/dL.
Diagnosed with lung cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) — Patient was diagnosed with lung cancer shortly after her 12 month study visit
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Constant Dose PTH (N=40) | Ascending Dose PTH (N=40)
Mild hypercalcemia or hypercalciuria (Endocrine disorders) | 3 (3) | 5 (5) — Asymptomatic
Joint pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (1) | 1 (1)
Lower extremity edema (Blood and lymphatic system disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No